CLINICAL TRIAL: NCT00062205
Title: Phase II Trial of Gleevec (STI571) in Therapy of Ewing's Family of Tumors and Desmoplastic Small Round Cell Tumors
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent Ewing's Family of Tumors or Desmoplastic Small Round-Cell Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Warren Chow MD, City of Hope Medical Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304551; P30CA033572 (NIH); CHNMC-IRB-02008
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Sarcoma
Keywords: recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: This phase II trial is studying how well imatinib mesylate works in treating patients with recurrent Ewing's family of tumors or desmoplastic small round-cell tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of imatinib mesylate in patients with recurrent Ewing's family of tumors or desmoplastic small round-cell tumor.
* Determine the toxic effects of this drug in these patients.
* Determine the duration of disease-free and overall survival of patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive oral imatinib mesylate twice daily on days 1-28. Courses repeat every 28 days.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Ewing's family of tumors OR desmoplastic small round-cell tumor
* Must have immunohistochemical evidence of expression of greater than 2+/4+ for either Kit (CD117) or platelet-derived growth factor receptor -a or -b
* No symptomatic brain metastases

  * Asymptomatic brain metastases are allowed provided patient is not on concurrent anticonvulsants or corticosteroids

PATIENT CHARACTERISTICS:

Age

* Over 16

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* No chronic active hepatitis
* No cirrhosis
* No other acute or known chronic liver disease

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No concurrent poorly controlled or severe cardiovascular disease

Pulmonary

* No concurrent poorly controlled or severe pulmonary disease

Other

* HIV negative
* No concurrent poorly controlled or severe central nervous system disease
* No other concurrent poorly controlled or severe nonmalignant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 3 weeks since prior chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* More than 2 weeks since prior major surgery

Other

* More than 28 days since prior investigational agents

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST criteria

SECONDARY OUTCOMES:
Progression-free survival at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States